CLINICAL TRIAL: NCT02663830
Title: The Effect of Sildenafil Citrate on the Success Rate of Ovulation Induction Using Clomiphene: A Randomized Controlled Trial.
Brief Title: The Effect of Sildenafil Citrate on the Success Rate of Ovulation Induction Using Clomiphene
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Ain Shams University (Other)
Responsible Party: Principal Investigator, Ahmed Abdel Shafy El Shahawy, Lecturer, Ain Shams University
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: SIOO
Record Dates: First submitted 2016-01-21; First posted 2016-01-26 (Estimated); Last update posted 2017-08-16 (Actual); Status verified 2017-08

CONDITIONS: Anovulatory
MeSH Terms: conditions — Anovulation | interventions — Sildenafil Citrate; Clomiphene

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- (Sildenafil & clomiphene citrate group) (Experimental): 105 Patients will receive 25 mg sildenafil citrate 6 hourly orally (day 6 to the end of the cycle), and clomiphene citrate 100 mg/day (day 2 to 6) orally by the patient, for induction of ovulation
  Interventions: Drug: Sildenafil & clomiphene citrate
- clomiphene only (Active Comparator): 105 patients will receive only clomiphene citrate 100mg/day (day 2 to 6) orally (2 tablets at same time daily).
  Interventions: Drug: clomiphene only

INTERVENTIONS:
Drug: Sildenafil & clomiphene citrate — 105 Patients will receive 25 mg sildenafil citrate 6hourly orally (day 6 to the end of the cycle), and clomiphene citrate 100 mg/day (day 2 to 6) orally by the patient, for induction of ovulation
  Other Names: seldin and clomid
  Arms: (Sildenafil & clomiphene citrate group)
Drug: clomiphene only — 105 Patients will receive clomiphene citrate 100 mg/day (day 2 to 6) orally by the patient, for induction of ovulation
  Other Names: clomid
  Arms: clomiphene only

SUMMARY:
The aim of the study is to evaluate the effect of sildenafil citrate on the pregnancy rate in women undergoing induction of ovulation using clomiphene citrate.

ELIGIBILITY:
Inclusion Criteria:

* Women age 21-35 years.
* Anovulatory cycles due to polycystic ovaries syndrome.
* Non-smokers.
* Free of major medical illness

Exclusion Criteria:

* Women with myoma or adenomyosis
* Women with congenital uterine anomaly.
* Chronic use of any medications including non-steroidal anti-inflammatory drugs.
* Associated cases of infertility other than PCOs (male factor, tubal factor,….).
* Asherman syndrome.
* Cases with endometrial hyperplasia.
* Cases with endometrial polyp

Ages: 21 Years to 35 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 210 (Actual)
Dates: Start 2016-01-10 (Actual); Primary Completion 2017-01-10 (Actual); Study Completion 2017-03-12 (Actual)

PRIMARY OUTCOMES:
Clinical pregnancy rate | 6 weeks

SECONDARY OUTCOMES:
endometrial thickness | 2 weeks
miscarriage rate | 13 weeks
ectopic pregnancy rate | 8 weeks
Side Effects of Vasodilators | 4 weeks

IPD SHARING:
Plan to Share IPD: Undecided